CLINICAL TRIAL: NCT04442594
Title: REMINISCENCES : Reminiscence Triggered by Virtual Reality for Older Adults With Mood Disorders
Brief Title: REMINISCENCES and EMOTIONS : Reminiscence Triggered by Virtual Reality for Older Adults With Mood Disorders
Acronym: REMINISCENCES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-PP-11
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease; Mood Disorders; Virtual Reality
MeSH Terms: conditions — Alzheimer Disease; Mood Disorders

STUDY DESIGN:
Intervention Model Description: The virtual reality sessions will take place twice a week during 6 weeks. Each subject will have two different virtual environment. The virtual environment will change every 3 weeks in order to avoid the phenomenon of habituation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized video (Experimental): Each subject of the reminiscence group will have two personalised virtual surroundings (after data being collected from team and/or families).
  Interventions: Procedure: virtual reality session
- generic vidéo (Active Comparator): The subjects of the control group will be exposed to two generic virtual settings (beach, mountain etc.)
  Interventions: Procedure: virtual reality session

INTERVENTIONS:
Procedure: virtual reality session — The virtual reality sessions will take place in a quiet setting twice a week in the living or hosting residence. The sessions will be hold over a period of time of 6 weeks.
  The virtual environment will change every 3 weeks in order to avoid the phenomenon of habituation.

SUMMARY:
Presentation & Pre-screening of the control group / reminiscence group Patient/resident pre-screening team meeting for the study Explanation and proposal of the study to patients and their families Signature of resident/patient and family consents Audit of inclusion and non-inclusion criteria Inclusion Medical advice for VR Clinical interview with the family or legal guardian for an accurate life history + an anamnesis interview (psychologist or doctor) with the patient or resident.

Creation of video contents Creation of personalized video contents Clinical scales review Evaluation of the number of psychotropic molecules prescribed (coordinating doctor, general practitioner, geriatrician)

* Pre-test phase with the patient for the use of the VR headset
* Randomisation
* Session procedure As previously mentioned, the virtual reality sessions will take place in a quiet setting twice a week in the living or hosting residence. The sessions will be hold over a period of time of 6 weeks.

Each subject of the reminiscence group will have two personalised virtual surroundings (after data being collected from team and/or families).

The virtual environment will change every 3 weeks in order to avoid the phenomenon of habituation.

The subjects of the control group will be exposed to two generic virtual settings (beach, mountain etc.) with a different virtual environment every 3 weeks.

During the session, note will be taken on the subject's speech. The session will also be filmed and/or recorded with a prior signed agreement by the patient or his representative.

- Last session (S6) Review of clinical scales (re-testing) Re-evaluation of drug prescriptions

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 65 or older
* Accompanied in day care or in the geriatric structure of the CHU of Nice (EHPAD-USLD)
* Mild to moderate cognitive impairment
* Diagnostic criteria for Alzheimer's disease, NINCDS-ADRDA probably,
* Positive score on at least one of the following rating scales :
* NPI-ES depression/dysphoria and anxiety items + GDS 15 Patients
* IA caregiver = 2 on one of 2 dimensions + IA patient = 2 on one of 2 dimensions

Exclusion Criteria:

* Diagnosed psychiatric pathology
* Disabling sensory disorders such as DMLA
* Significant hearing loss
* Subjects with risk of photosensitive epilepsy or dizziness. Subjects with Lewy body dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Depression and anxiety assessment | change of Hamilton score between inclusion and 6 weeks (before and after therapy)
  assessment with Hamilton scale

SECONDARY OUTCOMES:
psychotropic drugs consumption | change in psychotropic drugs consumption between inclusion and 6 weeks (before and after therapy)
  assessment of psychotropic drugs consumption

CONTACTS AND LOCATIONS:
Overall Officials: Olivier guerin.o@chu-nice.fr, PU-PH, Principal Investigator — Nice University Hospital, Gerontology Department
Locations (4):
- France (4):
  - CHU de Nice, Nice
  - EPHAD Ancilla, Nice
  - EPHAD Clos de Cimiez, Nice
  - Hopital privé Gériatrique Les Sources, Nice

IPD SHARING:
Plan to Share IPD: No